CLINICAL TRIAL: NCT01879696
Title: Double Blinded Study for the Reduction of the Incidence of Fasciotomy
Brief Title: Double Blinded, Randomized Clinical Trial of the Twin Star ECSPRESS Monitoring System for the Reduction of the Incidence of Fasciotomy
Acronym: ECSPRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Twin Star Medical, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-10000; G110163
Record Dates: First submitted 2013-06-11; First posted 2013-06-18 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Compartment Syndrome
MeSH Terms: conditions — Compartment Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Treatment are subjects will have catheter vacuum active for the removal of fluid from the muscle compartment.
  Interventions: Device: ECSPRESS catheter with active vacuum
- Control (No Intervention): Treatment are subjects will have catheter vacuum in-active for the removal of fluid from the muscle compartment.

INTERVENTIONS:
Device: ECSPRESS catheter with active vacuum
  Arms: Treatment

SUMMARY:
The proposed study is a double-blinded, randomized clinical trial of tissue pressure monitoring only (Control group) vs. tissue pressure monitoring plus tissue ultrafiltration (Treatment group) in patients with tibia fractures presenting to the trauma or emergency departments at participating clinical sites. Tissue ultrafiltration refers to the removal of muscle interstitial fluid by the ECSPRESS PMFC. The primary objective of the study is to demonstrate whether the removal of interstitial fluid by the ECSPRESS PMFC/FC catheters decrease the incidence of fasciotomy in the Treatment group when compared to the Control group. Fasciotomy was chosen as the primary outcome because it is clearly defined and clinically relevant; reduction of fasciotomy is of clear clinical benefit. Enrolled patients may have isolated tibia fractures OR be multiple trauma patients (those with another major fracture in a different body region or two distinct body system injuries, excluding those with injuries to the opposite leg that would preclude them from completing required tests).

DETAILED DESCRIPTION:
Eligible patients who are enrolled in the study will receive standard surgical stabilization within 72 hours of injury. All Subjects will receive the Twin Star ECSPRESS catheters, which will be inserted at the end of the surgical procedure to stabilize the tibia fracture and will be connected to the pressure monitor in the operating room or immediately upon arrival in the recovery room. The catheters will be used for up to 24-hours after surgical fixation of the affected lower leg in order to (1) measure and record muscle compartment pressure, and (2) remove interstitial fluid in the subset of subjects that are randomized to the Treatment Group. Subjects will be followed closely during the 24 hours the catheter is inserted to gather muscle pressure data, occurrance of a fasciotomy, adverse events, etc. and then followed up at 2 weeks, 3 months, 6 months and 12 months post study enrollment after which the subjects participation in the study will be completed. There will no interim data analysis of the study outcomes during the conduct of this study. Data analysis and presentation of the data will be made after study closure.

ELIGIBILITY:
Inclusion Criteria:

* • Subject with an isolated tibial shaft fracture requiring intramedullary nailing, or bicondylar tibial plateau fracture or tibial plateau fracture-knee dislocation requiring application of a knee-spanning external fixator. OR Subject with an isolated tibial shaft fracture requiring intramedullary nailing, or bicondylar tibial plateau fracture or tibial plateau fracture-knee dislocation requiring application of a knee-spanning external fixator AND another major fracture in a different body region or injuries to one other major organ system (head, chest, abdomen, pelvis, genitourinary, or spine) excluding those with injuries to the opposite leg that would preclude them from completing required tests (see exclusion criteria).
* • Subject with an isolated tibial shaft fracture requiring intramedullary nailing, or bicondylar tibial plateau fracture or tibial plateau fracture-knee dislocation requiring application of a knee-spanning external fixator AND another major fracture in a different body region or injuries to one other major organ system (head, chest, abdomen, pelvis, genitourinary, or spine) excluding those with injuries to the opposite leg that would preclude them from completing required tests (see exclusion criteria).

All Subjects

* Operative procedure (nailing or external fixation) performed within 72 hours of injury.
* The Subject is at least 18 years of age and no older than 44 years of age. Subject or legally acceptable representative must able to understand what he/she is being asked to do, willing/able to understand and sign the Informed Consent to return for the required follow-up visits at 2 weeks, 3 months, 6 months, and 12 months post-surgery. A legally acceptable representative may sign the Informed Consent on the patient's behalf.
* In the study investigators opinion, patient's co-morbidity condition(s) at enrollment WILL allow patient to return and complete the required testing for all return visits for the duration of this 12-month clinical study.

Exclusion Criteria:

* • Current evidence of CS prior to the decision regarding enrollment. Surgical stabilization that resulted in the presence of a bead pouch, VAC, negative-pressure wound therapy device, or other dressing that would interfere with placement of any of the four catheters in the anterior deep posterior compartments.

  * The Subject has a medical condition(s) that precludes use of catheters, such as dermatologic conditions, immunological deficits, or traumatic skin lesions that interfere with Catheter placement.
  * An Injury to the ipsilateral knee, ankle, and/or foot that would influence results of muscle testing.
  * Opposite leg knee injury or tibia, ankle, foot fracture, or any other injury that would preclude or influence the results of mechanical muscle testing.
  * Incision into the anterior or deep posterior compartments of the leg to be studied that would release the fascia as this would constitute a partial fasciotomy and would affect leg pressures.
  * The Subject is currently enrolled in one or more clinical studies.
  * Likely problems, in the investigator's judgment, with maintaining follow-up (including developmental delay, address greater than 2 hours drive from the treating institution, substance abuse problems, intoxication, current or pending incarceration, etc.).

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of fasciotomies | End of study once all subjects have completed their 12 month follow-up interval.

SECONDARY OUTCOMES:
Area under the curve (AUC) for time-pressure | End of study once all subjects have completed their 12 month follow-up interval.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States